CLINICAL TRIAL: NCT02472795
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-response Study to Investigate the Biological Activity, Safety, Tolerability, and Pharmacokinetics of ACT-334441 in Subjects With Systemic Lupus Erythematosus
Brief Title: Clinical Study to Investigate the Biological Activity, Safety, Tolerability, and Pharmacokinetics of ACT-334441 in Subjects With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-064A201
Record Dates: First submitted 2015-05-14; First posted 2015-06-16 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2020-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — cenerimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cenerimod 0.5 mg (Part A) (Experimental): Participants will receive cenerimod 0.5 mg capsules orally once daily for 12 weeks.
  Interventions: Drug: Cenerimod
- Cenerimod 1 mg (Part A) (Experimental): Participants will receive cenerimod 1 mg capsules orally once daily for 12 weeks.
  Interventions: Drug: Cenerimod
- Cenerimod 2 mg (Part A) (Experimental): Participants will receive cenerimod 2 mg capsules orally once daily for 12 weeks.
  Interventions: Drug: Cenerimod
- Cenerimod 4 mg (Part B) (Experimental): Participants will received cenerimod 4 mg capsules orally once daily for 12 weeks. This treatment arm will start after all patients in Part A have completed 4 weeks of placebo, 0.5 mg, 1 mg and 2 mg cenerimod treatment.
  Interventions: Drug: Cenerimod
- Matching placebo (Part A and B) (Placebo Comparator): Capsules of matching placebo taken orally once daily for 12 weeks.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Matching placebo — One capsule of cenerimod to be taken once daily, irrespective of food intake. The capsule is to be swallowed whole. The capsule should be taken each day at approximately the same time (preferably each morning).
  Other Names: Placebo
  Arms: Matching placebo (Part A and B)
Drug: Cenerimod — One capsule of cenerimod to be taken once daily, irrespective of food intake. The capsule is to be swallowed whole. The capsule should be taken each day at approximately the same time (preferably each morning).
  Other Names: ACT-334441
  Arms: Cenerimod 0.5 mg (Part A); Cenerimod 1 mg (Part A); Cenerimod 2 mg (Part A); Cenerimod 4 mg (Part B)

SUMMARY:
International trial to evaluate the biological activity and safety of cenerimod (ACT-334441) in systemic lupus erythematosus (SLE) patients.

DETAILED DESCRIPTION:
This multicentre, double-blind, placebo-controlled study will have a staggered approach (Part A and B).

In part A, eligible patients will be randomly assigned (1:1:1:1) to once daily oral administration of cenerimod (0.5, 1, 2 mg) or placebo. After all patients have completed 4 weeks of treatment during part A, an Independent Data Monitoring Committee will review non-blinded data in an interim analysis to evaluate the safety profile of cenerimod and recommend whether the study could proceed to part B.

In part B, additional patients will be randomized (3:1) to once daily oral administration of cenerimod 4 mg or placebo.

All participants will receive study medication for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 to 65 years with established SLE. Participants must have active SLE, Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) score of at least 2 points for musculoskeletal or mucocutaneous manifestations and history or presence at screening of positive anti-nuclear antibodies (ANA) or anti-double-stranded DNA (anti-dsDNA) antibodies.
* Enrolled participants must be treated with background SLE medications.

Exclusion Criteria:

* Participants with significant medical conditions or therapies for such conditions (e.g., cardiovascular, pulmonary, immunological, hepatic, ophthalmological, infection and infection risks, history or presence of malignancy, history or presence of bone marrow or solid organ transplantation) or lactating or pregnant women.
* Participants with severe SLE disease or with clinically relevant medical or surgical conditions that, in the opinion of the investigator, would put the subject at risk by participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (15):
- United States (2):
  - Investigator Site, Anniston, Alabama
  - Investigator Site, Clearwater, Florida
- Belarus (2):
  - Investigator Site, Minsk
  - Investigator Site, Vitebsk
- Bulgaria (2):
  - Investigator Site, Plovdiv
  - Investigator Site, Sofia
- Investigator Site, Tbilisi, Georgia
- Russia (6):
  - Investigator Site, Kemerovo
  - Investigator Site, Kursk
  - Investigator Site, Omsk
  - Investigator Site, Orenburg
  - Investigator Site, Smolensk
  - Investigator Site, Vladimir
- Ukraine (2):
  - Investigator Site, Vinnytsia
  - Investigator Site, Zaporizhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hermann V, Batalov A, Smakotina S, Juif PE, Cornelisse P. First use of cenerimod, a selective S1P1 receptor modulator, for the treatment of SLE: a double-blind, randomised, placebo-controlled, proof-of-concept study. Lupus Sci Med. 2019 Nov 9;6(1):e000354. doi: 10.1136/lupus-2019-000354. eCollection 2019. PMID 31798918
- See also: Lay summary on results reference by Hermann V et al. First use of cenerimod, a selective S1P(1) receptor modulator, for the treatment of SLE: a double-blind, randomised, placebo-controlled, proof-of-concept study. Lupus Sci Med. 2019 Nov 9;6(1):e000354. — https://lupus.bmj.com/content/lupusscimed/suppl/2019/11/12/6.1.e000354.DC4/lupus-2019-000354_lay_summary.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 18 sites in 6 countries between 1 June 2015 and 28 February 2017, 105 patients signed consent and 67 were randomized to a study treatment: 49 in part A (randomized 1:1:1:1 to receive cenerimod 0.5, 1, 2 mg or placebo) and 18 in part B (randomized 3:1 to receive cenerimod 4 mg or placebo).
Pre-assignment Details: The screening period started when the informed consent was signed (up to 30 days before randomization), and ended with randomization. The period included Visit 1 (screening) and the pre-randomization (pre-dose) assessments at Visit 2 (Day 1). Thirty-two patients did not meet the inclusion/exclusion criteria and 6 patients withdrew from the study.
Groups:
- Cenerimod 0.5 mg (Part A): Participants received cenerimod 0.5 mg capsules orally once daily for 12 weeks.
- Cenerimod 1 mg (Part A): Participants received cenerimod 1 mg capsules orally once daily for 12 weeks.
- Cenerimod 2 mg (Part A): Participants received cenerimod 2 mg capsules orally once daily for 12 weeks.
- Cenerimod 4 mg (Part B): Participants received cenerimod 4 mg capsules orally once daily for 12 weeks.
- Matching Placebo (Part A and B): Participants received cenerimod matching placebo capsules orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Cenerimod 0.5 mg (Part A) | Cenerimod 1 mg (Part A) | Cenerimod 2 mg (Part A) | Cenerimod 4 mg (Part B) | Matching Placebo (Part A and B)
Started | 12 | 12 | 13 | 13 | 17
Pharmacodynamic Set | 12 | 10 | 13 | 13 | 16
Modified Pharmacodynamic Analysis Set | 12 | 10 | 13 | 9 | 16
Completed | 12 | 11 | 13 | 13 | 14
Not Completed | 0 | 1 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (N=67). Pharmacodynamic analysis set (PD set, N=64) at least 21 days of treatment, with lymphocyte count measurements at baseline and post-baseline.
  Modified pharmacodynamic analysis set (N=60) excluded 4 patients from PD set with low, or below the lower limit of quantification (BLQ) Ctrough levels.
Groups:
- Matching Placebo (Part A and Part B): Participants received cenerimod matching placebo capsules orally once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Cenerimod 0.5 mg (Part A) | Cenerimod 1 mg (Part A) | Cenerimod 2 mg (Part A) | Cenerimod 4 mg (Part B) | Matching Placebo (Part A and Part B) | Total
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 17 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Different population analysis sets.
  years
    Full analysis set | 41.4 (13.2) | 37.0 (6.4) | 39.2 (11.8) | 41.7 (8.1) | 41.0 (9.5) | 40.1 (9.9)
    Pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 13 | 16 | 64
    Pharmacodynamic analysis set | 41.4 (13.2) | 38.1 (5.4) | 39.2 (11.8) | 41.7 (8.1) | 41.8 (9.2) | 40.6 (9.8)
    Modified pharmacodynamics analysis set: number analyzed (Participants) | 12 | 10 | 13 | 9 | 16 | 60
    Modified pharmacodynamics analysis set | 41.4 (13.2) | 38.1 (5.4) | 39.2 (11.8) | 41.9 (8.6) | 41.8 (9.2) | 40.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Different population analysis sets.
  Participants
    Full analysis set: Female | 11 | 12 | 12 | 10 | 16 | 61
    Full analysis set: Male | 1 | 0 | 1 | 3 | 1 | 6
    Pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 13 | 16 | 64
    Pharmacodynamic analysis set: Female | 11 | 10 | 12 | 10 | 16 | 59
    Pharmacodynamic analysis set: Male | 1 | 0 | 1 | 3 | 0 | 5
    Modified pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 9 | 16 | 60
    Modified pharmacodynamic analysis set: Female | 11 | 10 | 12 | 7 | 16 | 56
    Modified pharmacodynamic analysis set: Male | 1 | 0 | 1 | 2 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 13 | 13 | 17 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Different population analysis sets.
  Participants
    Full analysis set: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Full analysis set: Asian | 0 | 0 | 0 | 0 | 0 | 0
    Full analysis set: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Full analysis set: Black or African American | 0 | 0 | 0 | 0 | 2 | 2
    Full analysis set: White | 12 | 12 | 13 | 13 | 15 | 65
    Full analysis set: More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Full analysis set: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
    Pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 13 | 16 | 64
    Pharmacodynamic analysis set: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Pharmacodynamic analysis set: Asian | 0 | 0 | 0 | 0 | 0 | 0
    Pharmacodynamic analysis set: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Pharmacodynamic analysis set: Black or African American | 0 | 0 | 0 | 0 | 2 | 2
    Pharmacodynamic analysis set: White | 12 | 10 | 13 | 13 | 14 | 62
    Pharmacodynamic analysis set: More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Pharmacodynamic analysis set: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
    Modified pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 9 | 16 | 60
    Modified pharmacodynamic analysis set: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Modified pharmacodynamic analysis set: Asian | 0 | 0 | 0 | 0 | 0 | 0
    Modified pharmacodynamic analysis set: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Modified pharmacodynamic analysis set: Black or African American | 0 | 0 | 0 | 0 | 2 | 2
    Modified pharmacodynamic analysis set: White | 12 | 10 | 13 | 9 | 14 | 58
    Modified pharmacodynamic analysis set: More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Modified pharmacodynamic analysis set: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 0 | 0 | 2 | 4
  Ukraine | 3 | 1 | 2 | 1 | 2 | 9
  Georgia | 2 | 1 | 1 | 1 | 1 | 6
  Belarus | 0 | 1 | 2 | 2 | 2 | 7
  Bulgaria | 3 | 2 | 2 | 7 | 5 | 19
  Russia | 3 | 6 | 6 | 2 | 5 | 22
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: Different population analysis sets.
  kg/m^2
    Full analysis set | 25.2 (5.1) | 27.4 (8.0) | 26.0 (5.1) | 27.5 (4.7) | 25.4 (6.8) | 26.3 (6.0)
    Pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 13 | 16 | 64
    Pharmacodynamic analysis set | 25.2 (5.1) | 28.8 (8.1) | 26.0 (5.1) | 27.5 (4.7) | 25.5 (7.0) | 26.5 (6.1)
    Modified pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 9 | 16 | 60
    Modified pharmacodynamic analysis set | 25.2 (5.1) | 28.8 (8.1) | 26.0 (5.1) | 28.3 (5.4) | 25.5 (7.0) | 26.5 (6.2)
Disease history time from first Systemic Lupus Erythematosus symptoms [Median (Full Range); unit: years] — Population: Different population analysis sets.
  years
    Full analysis set | 3.7 [1.6 to 23.7] | 8.2 [0.6 to 22.5] | 6.7 [1.4 to 20.9] | 4.6 [0.8 to 10.5] | 7.9 [1.1 to 22.1] | 6.0 [0.6 to 23.7]
    Pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 13 | 16 | 64
    Pharmacodynamic analysis set | 3.7 [1.6 to 23.7] | 9.2 [0.6 to 22.5] | 6.7 [1.4 to 20.9] | 4.6 [0.8 to 10.5] | 7.9 [1.7 to 22.1] | 6.2 [0.6 to 23.7]
    Modified pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 9 | 16 | 60
    Modified pharmacodynamic analysis set | 3.7 [1.6 to 23.7] | 9.2 [0.6 to 22.5] | 6.7 [1.4 to 20.9] | 3.2 [0.8 to 6.7] | 7.9 [1.7 to 22.1] | 6.2 [0.6 to 23.7]
Time from first Systemic Lupus Erythematosus diagnosis [Median (Full Range); unit: years] — Population: Different population analysis sets.
  years
    Full analysis set | 2.4 [1.4 to 23.7] | 6.2 [0.5 to 22.3] | 4.5 [1.3 to 17.0] | 2.9 [0.6 to 9.2] | 4.9 [0.5 to 21.4] | 3.8 [0.5 to 23.7]
    Pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 13 | 16 | 64
    Pharmacodynamic analysis set | 2.4 [1.4 to 23.7] | 5.8 [0.5 to 22.3] | 4.5 [1.3 to 17.0] | 2.9 [0.6 to 9.2] | 5.0 [0.5 to 21.4] | 3.6 [0.5 to 23.7]
    Modified pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 9 | 16 | 60
    Modified pharmacodynamic analysis set | 2.4 [1.4 to 23.7] | 5.8 [0.5 to 22.3] | 4.5 [1.3 to 17.0] | 1.3 [0.6 to 5.2] | 5.0 [0.5 to 21.4] | 3.6 [0.5 to 23.7]
Number of American College of Rheumatology criteria ongoing at screening [Count of Participants; unit: Participants] — The American College of Rheumatology (ACR) has designated 11 classification criteria incorporating major clinical features (mucocutaneous, articular, serosal, renal, and neurologic) and laboratory findings (hematologic and immunologic), which have been validated for the diagnosis of SLE. The presence of 4 or more criteria occurring either simultaneously or in succession is strongly suggestive of the diagnosis of SLE [Hochberg MC. Updating the American College of Rheumatology revised criteria for the classification of systemic lupus erythematosus. Arthritis Rheum 1997;40(9).]
  Participants
    0 to 3 ACR criteria ongoing at screening | 5 | 3 | 5 | 1 | 6 | 20
    4 to 11 ACR criteria ongoing at screening | 7 | 9 | 8 | 12 | 11 | 47
    0 to 3 ACR criteria more than 6 months ago | 0 | 0 | 0 | 0 | 0 | 0
    4 to 11 ACR criteria more than 6 months ago | 12 | 12 | 13 | 13 | 17 | 67
Systemic Lupus Erythematosus Disease Activity Index-2000, modified to exclude leucopenia [Mean (Standard Deviation); unit: units on a scale] — The SLEDAI-2K is a weighted, cumulative index of lupus disease activity scored by the physician. It is calculated from 24 individual descriptors across 9 organ systems, 0 indicates inactive disease and the maximum theoretical score is 105 (Gladman D et al. J Rheumatol 2002;29;288-291). In this study the SLEDAI-2K was modified, to exclude leucopenia (1 point), due to the mechanism of action of cenerimod. A score of 6 or greater is clinically relevant and associated with requiring lupus-directed therapy (Nuttall A et al. Best Pract Res Clin Rheumatol. 2013 Jun; 27(3):309-18). Population: Different population analysis sets.
  units on a scale
    Full analysis set | 7.3 (3.3) | 8.3 (3.7) | 7.1 (2.3) | 8.7 (3.1) | 7.4 (3.3) | 7.7 (3.1)
    Pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 13 | 16 | 64
    Pharmacodynamic analysis set | 7.3 (3.3) | 7.0 (2.2) | 7.1 (2.3) | 8.7 (3.1) | 7.3 (3.4) | 7.5 (2.9)
    Modified pharmacodynamic analysis set: number analyzed (Participants) | 12 | 10 | 13 | 9 | 16 | 60
    Modified pharmacodynamic analysis set | 7.3 (3.3) | 7.0 (2.2) | 7.1 (2.3) | 8.1 (2.5) | 7.3 (3.4) | 7.3 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Lymphocyte Count From Baseline to End-of-treatment (EOT)
Description: The primary objective of the clinical study was to asses whether cenerimod could reduce the number of circulating lymphocytes in the bloodstream of people with systemic lupus erythematosus (SLE).
  The change was defined as: Total lymphocyte count at end-of-treatment (EOT) minus total lymphocyte count at baseline.
  A negative change over time indicates that the number of peripheral circulating lymphocytes has decreased.
  The reduction of the total lymphocyte count over a treatment period indicates a pharmacodynamic effect.
  The value at baseline was defined as the last non-missing value obtained from a sample taken prior to the first study treatment intake.
  End-of-treatment (EOT) was defined as the last post-baseline value with treatment for at least 21 days up to Week 12.
Time Frame: Baseline to end-of-treatment (EOT) (up to 12 weeks)
Population: Pharmacodynamics analysis (PD) set. The PD set includes all participants who received at least 21 days of study treatment, with lymphocyte count measurements at baseline and post-baseline. Last observation carried forward (using the Week 4 visit or later) was used for participants with a missing end-of-treatment (EOT) assessment.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Groups:
- Matching Placebo: Participants received cenerimod matching placebo capsules orally once daily for 12 weeks.
Arm/Group | Cenerimod 0.5 mg (Part A) | Cenerimod 1 mg (Part A) | Cenerimod 2 mg (Part A) | Cenerimod 4 mg (Part B) | Matching Placebo
Number analyzed (Participants) | 12 | 10 | 13 | 13 | 16
10^9 cells/L | -0.26 (0.48) | -0.96 (0.68) | -0.86 (0.61) | -0.87 (1.24) | -0.33 (0.72)
Statistical Analysis 1: Comparison: Cenerimod 0.5 mg (Part A) vs Matching Placebo; Test type: Superiority; p = 0.39, ANCOVA; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.56 to 0.22], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Cenerimod 1 mg (Part A) vs Matching Placebo; Test type: Superiority; p = 0.02, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.91 to 0.09], Standard Error of Mean 0.2
Statistical Analysis 3: Comparison: Cenerimod 2 mg (Part A) vs Matching Placebo; Test type: Superiority; p = 0.004, ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.95 to -0.19], Standard Error of Mean 0.19
Statistical Analysis 4: Comparison: Cenerimod 4 mg (Part B) vs Matching Placebo; Test type: Superiority; p = 0.06, ANCOVA; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.75 to 0.02], Standard Error of Mean 0.19

2. Primary Outcome: Change in Total Lymphocyte Count From Baseline to Each Post-baseline Assessment
Description: The primary objective of the clinical study was to assess whether cenerimod could reduce the number of circulating lymphocytes in the bloodstream of people with systemic lupus erythematosus (SLE).
  The change was defined as: Total lymphocyte count at visit minus total lymphocyte count at baseline.
  A negative change over time indicates that the number of peripheral circulating lymphocytes has decreased.
  The reduction of the total lymphocyte count over a treatment period indicates a pharmacodynamic effect.
  The value at baseline was defined as the last non-missing value obtained from a sample taken prior to the first study treatment intake.
  End-of-treatment (EOT) was defined as the last post-baseline value with treatment for at least 21 days up to Week 12.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, end-of-treatment Visit (up to 12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Cenerimod 0.5 mg (Part A) | Cenerimod 1 mg (Part A) | Cenerimod 2 mg (Part A) | Cenerimod 4 mg (Part B) | Matching Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 17
10^9 cells/L
  Baseline visit | 1.37 (0.52) | 1.71 (0.82) | 1.62 (0.75) | 1.88 (0.77) | 1.65 (0.88)
  Week 2 visit: number analyzed (Participants) | 12 | 8 | 12 | 13 | 16
  Week 2 visit | -0.13 (0.56) | -0.48 (0.56) | -0.52 (1.03) | -1.09 (0.65) | -0.16 (0.75)
  Week 4 visit: number analyzed (Participants) | 12 | 11 | 12 | 13 | 16
  Week 4 visit | -0.28 (0.42) | -0.69 (0.76) | -0.86 (0.63) | -0.68 (1.32) | -0.33 (0.69)
  Week 8 Visit: number analyzed (Participants) | 12 | 10 | 13 | 13 | 14
  Week 8 Visit | -0.28 (0.60) | -0.92 (0.60) | -0.89 (0.68) | -1.03 (1.12) | -0.09 (0.82)
  Week 12 visit: number analyzed (Participants) | 12 | 11 | 13 | 13 | 13
  Week 12 visit | -0.26 (0.48) | -0.72 (1.03) | -0.86 (0.61) | -0.87 (1.24) | -0.29 (0.73)
  End-of-treatment visit: number analyzed (Participants) | 12 | 11 | 13 | 13 | 17
  End-of-treatment visit | -0.26 (0.48) | -0.72 (1.03) | -0.86 (0.61) | -0.87 (1.24) | -0.30 (0.71)

3. Post Hoc Outcome: Change in Total Lymphocyte Count From Baseline to End-of-treatment (EOT) Based on Pharmacokinetic Cthrough Profiles
Description: The change was defined as: Total lymphocyte count at end-of-treatment (EOT) minus total lymphocyte count at baseline.
  A negative change over time indicates that the number of peripheral circulating lymphocytes has decreased.
  The value at baseline was defined as the last non-missing value obtained from a sample taken prior to the first study treatment intake.
  End-of-treatment (EOT) was defined as the last post-baseline value with treatment for at least 21 days up to Week 12.
  The modified pharmacodynamics analysis set includes all participants who:
  * received at least 21 days of study treatment &
  * with lymphocyte count measurements at baseline and post-baseline (namely, one sample taken at least 21 days after the first study treatment intake and no later than 7 days after the last study treatment intake with no treatment interruption documented in the first 21 days) &
  * with cenerimod plasma concentrations at Week 4 consistent with expectations.
Time Frame: Baseline to end-of-treatment (EOT) (up to 12 weeks)
Population: Ctrough levels were discovered to be low, or below the lower limit of quantification (BLQ), in four patients randomized to the cenerimod 4 mg group, a finding incompatible with compliance with study treatment. These patients were excluded from the pharmacodynamic analysis set to form a modified pharmacodynamics analysis set.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Cenerimod 0.5 mg (Part A) | Cenerimod 1 mg (Part A) | Cenerimod 2 mg (Part A) | Cenerimod 4 mg (Part B) | Matching Placebo
Number analyzed (Participants) | 12 | 10 | 13 | 9 | 16
10^9 cells/L | -0.26 (0.48) | -0.96 (0.68) | -0.86 (0.61) | -1.48 (0.73) | -0.32 (0.72)
Statistical Analysis 1: Comparison: Cenerimod 0.5 mg (Part A) vs Matching Placebo; Test type: Superiority; p = 0.2837, ANCOVA; Mean Difference (Final Values) = -0.145, 95% CI 2-sided [-0.413 to 0.123], Standard Error of Mean 0.134
Statistical Analysis 2: Comparison: Cenerimod 1 mg (Part A) vs Matching Placebo; Test type: Superiority; p = 0.0006, ANCOVA; Mean Difference (Final Values) = -0.515, 95% CI 2-sided [-0.797 to -0.234], Standard Error of Mean 0.140
Statistical Analysis 3: Comparison: Cenerimod 2 mg (Part A) vs Matching Placebo; Test type: Superiority; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -0.565, 95% CI 2-sided [-0.825 to -0.305], Standard Error of Mean 0.130
Statistical Analysis 4: Comparison: Cenerimod 4 mg (Part B) vs Matching Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.880, 95% CI 2-sided [-1.173 to -0.586], Standard Error of Mean 0.147

4. Post Hoc Outcome: Absolute Values of Total Lymphocyte Count at Each Analysis Visit
Description: The primary objective of the clinical study was to see whether cenerimod could reduce the number of circulating lymphocytes in the bloodstream of people with systemic lupus erythematosus (SLE).
  The reduction of the total lymphocyte count over a treatment period indicates a pharmacodynamic effect.
  The modified pharmacodynamics analysis set includes all participants who:
  * received at least 21 days of study treatment &
  * with lymphocyte count measurements at baseline and post-baseline (namely, one sample taken at least 21 days after the first study treatment intake and no later than 7 days after the last study treatment intake with no treatment interruption documented in the first 21 days) &
  * with cenerimod plasma concentrations at Week 4 consistent with expectations.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, end-of-treatment (EOT - up to 12 weeks), end-of-study (6 weeks after EOT)
Population: All participants for which data was available. Ctrough levels were discovered to be low, or below the lower limit of quantification (BLQ), in four patients randomised to the cenerimod 4 mg group, a finding incompatible with compliance with study treatment. These patients were excluded from the PD set to form a modified pharmacodynamic analysis set.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Cenerimod 0.5 mg (Part A) | Cenerimod 1 mg (Part A) | Cenerimod 2 mg (Part A) | Cenerimod 4 mg (Part B) | Matching Placebo
Number analyzed (Participants) | 12 | 10 | 13 | 9 | 16
10^9 cells/L
  Baseline visit | 1.37 (0.52) | 1.83 (0.79) | 1.62 (0.75) | 2.04 (0.80) | 1.66 (0.91)
  Week 2 visit: number analyzed (Participants) | 12 | 8 | 12 | 9 | 15
  Week 2 visit | 1.24 (0.34) | 1.38 (0.49) | 1.19 (0.89) | 0.79 (0.44) | 1.44 (0.44)
  Week 4 visit: number analyzed (Participants) | 12 | 10 | 12 | 9 | 15
  Week 4 visit | 1.09 (0.27) | 0.99 (0.38) | 0.73 (0.39) | 0.71 (0.49) | 1.31 (0.5)
  Week 8 visit: number analyzed (Participants) | 12 | 10 | 13 | 9 | 13
  Week 8 visit | 1.08 (0.43) | 0.91 (0.40) | 0.73 (0.36) | 0.51 (0.28) | 1.49 (0.73)
  Week 12 visit | 1.11 (0.37) | 0.87 (0.34) | 0.76 (0.44) | 0.57 (0.21) | 1.33 (0.54)
  End-of-treatment visit | 1.11 (0.37) | 0.87 (0.34) | 0.76 (0.44) | 0.57 (0.21) | 1.34 (0.51)
  End-of-study visit | 1.42 (0.37) | 1.42 (0.58) | 1.35 (0.45) | 1.14 (0.52) | 1.71 (0.86)

5. Post Hoc Outcome: Total Lymphocyte Count Percent Change From Baseline to End-of-treatment (EOT)
Description: Percentage change in total lymphocyte count from baseline to end-of-treatment (EOT).
  Percent change from baseline is defined as the absolute change from baseline divided by the baseline value (if the baseline value is > 0) and then multiplied by 100.
  A negative change over time indicates that the number of peripheral circulating lymphocytes has decreased.
  The reduction of the total lymphocyte count over a treatment period indicates a pharmacodynamic effect.
  The modified pharmacodynamics analysis set includes all participants who:
  * received at least 21 days of study treatment &
  * with lymphocyte count measurements at baseline and post-baseline (namely, one sample taken at least 21 days after the first study treatment intake and no later than 7 days after the last study treatment intake with no treatment interruption documented in the first 21 days) &
  * with cenerimod plasma concentrations at Week 4 consistent with expectations.
Time Frame: Baseline to End of Treatment (EOT) (up to 12 weeks)
Population: Ctrough levels were discovered to be low, or below the lower limit of quantification (BLQ), in four patients randomized to the cenerimod 4 mg group, a finding incompatible with compliance with study treatment. These patients were excluded from the pharmacodynamic set to form a modified pharmacodynamic analysis set.
Measure: Mean (Standard Deviation); unit: Percent change of total lymphocyte count
Arm/Group | Cenerimod 0.5 mg (Part A) | Cenerimod 1 mg (Part A) | Cenerimod 2 mg (Part A) | Cenerimod 4 mg (Part B) | Matching Placebo
Number analyzed (Participants) | 12 | 10 | 13 | 9 | 16
Percent change of total lymphocyte count | -12.23 (34.29) | -47.76 (20.37) | -51.52 (22.53) | -69.27 (13.68) | -5.04 (39.22)
Statistical Analysis 1: Comparison: Cenerimod 0.5 mg (Part A) vs Matching Placebo; Test type: Superiority; p = 0.1755, ANCOVA; Mean Difference (Final Values) = -13.214, 95% CI 2-sided [-32.513 to 6.085], Standard Error of Mean 9.626
Statistical Analysis 2: Comparison: Cenerimod 1 mg (Part A) vs Matching Placebo; Test type: Superiority; p = 0.0003, ANCOVA; Mean Difference (Final Values) = -39.311, 95% CI 2-sided [-59.552 to -19.069], Standard Error of Mean 10.096
Statistical Analysis 3: Comparison: Cenerimod 2 mg (Part A) vs Matching Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -47.278, 95% CI 2-sided [-65.981 to -28.574], Standard Error of Mean 9.329
Statistical Analysis 4: Comparison: Cenerimod 4 mg (Part B) vs Matching Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -56.452, 95% CI 2-sided [-77.585 to -35.320], Standard Error of Mean 10.541

ADVERSE EVENTS:
Time Frame: All Adverse Events and Serious Adverse Events that occurred after the intake of the first study treatment and up to 6 weeks after study treatment discontinuation are reported, assessed up to 18 weeks.
Groups:
- Cenerimod 0.5 mg: Participants received cenerimod 0.5 mg capsules orally once daily for 12 weeks.
- Cenerimod 1 mg: Participants received cenerimod 1 mg capsules orally once daily for 12 weeks.
- Cenerimod 2 mg: Participants received cenerimod 2 mg capsules orally once daily for 12 weeks.
- Cenerimod 4 mg: Participants received cenerimod 4 mg capsules orally once daily for 12 weeks.
Arm/Group | Cenerimod 0.5 mg | Cenerimod 1 mg | Cenerimod 2 mg | Cenerimod 4 mg | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13 | 1/17
Other Adverse Events (participants affected / at risk) | 5/12 | 5/12 | 6/13 | 5/13 | 9/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cenerimod 0.5 mg (N=12) | Cenerimod 1 mg (N=12) | Cenerimod 2 mg (N=13) | Cenerimod 4 mg (N=13) | Matching Placebo (N=17)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cenerimod 0.5 mg (N=12) | Cenerimod 1 mg (N=12) | Cenerimod 2 mg (N=13) | Cenerimod 4 mg (N=13) | Matching Placebo (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T wave amplitude decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nitrituria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study is the first to investigate short-term cenerimod treatment in patients with mild to moderate systemic lupus erythematosus (SLE).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT02472795/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT02472795/SAP_001.pdf